CLINICAL TRIAL: NCT03034798
Title: The Effects of Basal Insulin Suspension at the Start of Exercise on Blood Glucose Levels During Continuous vs. Circuit-based Exercise in Individuals With Type 1 Diabetes on CSII
Brief Title: Suspending Basal Insulin Levels for Exercise in Adults With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: York University (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Principal Investigator, Michael Riddell, Professor, York University
Other Study IDs: 1DP3DK101075 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Type1 Diabetes Mellitus; Physical Activity; Hypoglycemia
MeSH Terms: conditions — Motor Activity; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 Diabetes Exercisers: Participants performed 2 different forms of exercise of identical duration and similar total energy expenditure. One form was purely aerobic in nature and the other was intermittent, high-intensity exercise.

SUMMARY:
The purpose of the study is to determine the effects of insulin suspension at start of exercise in individuals with type 1 diabetes. A total of 3 sessions will be required for this project. The first will be a familiarization session that requires completed informed consent, anthropometric measurements (height, weight, body fat percentage), questionnaires, and a test of maximal aerobic fitness. The remaining 2 sessions will be steady-state aerobic exercise as well as circuit exercise.

DETAILED DESCRIPTION:
Written informed consent will be collected on the first day during the familiarization session from all individuals that wish to participate. A researcher will provide a brief explanation on how the continuous glucose monitor (CGM) works (Medtronic Inc., Canada) during the first visit to the laboratory. They will also describe how the CGM sensor insertion process will occur for those participants who have not worn one in the past. The participant will clean and sanitize the area and insert the CGM superficially in the skin themselves and connect the transmitter device to the sensor. The CGM will be worn for a total of 7 days and then removed by the participant and returned to the researcher to be downloaded. The sports armband will also be placed on the left upper arm and be worn continuously for 7 days. The principal student investigator (PSI) or principal investigator (PI) will provide all participants with information about the sports armband and place it on the skin immediately following. This device simply sits on the surface of the skin, but has a specific placement and activation and must be applied by the PSI or PI. Finally, during exercise visits, the Zephyr bioharness will be connected just below chest level and around the rib cage. This device is sits on top of the skin simply like an elastic band around the rib cage. The bioharness will only be worn during exercise visits and disconnected at the end of each activity.

Blood glucose levels will be monitored frequently during exercise using a Contour Link glucometer (Bayer, Canada). Participants will use personal lancing device for finger pokes, but the investigators will provide the glucometer and test strips. Each blood sugar check will be recorded in the data binder along with carbohydrate intake, any changes in basal rate or pump settings, and food intake. If blood glucose levels reach 3.9 mmol/L or less, participants will be asked to stop activity immediately and consume fast-acting carbohydrates (i.e. Dextrose tablets (Dex4, USA)). 15-minutes after ingestion of carbohydrates, blood glucose will be tested again before allowing the individual to return to activity safely. On the last day of testing, participants will be asked to return the CGM, sports armband, and bioharness to the research team. The data will later be uploaded and analyzed.

Patients will undergo a fitness assessment (maximal aerobic capacity) during visit 1 and perform 40-minutes of continuous (treadmill jogging) and 40-minutes of intermittent (calisthenics) high-intensity type exercises (visit 2 and 3). Upon entry to the laboratory, participants will be asked to check blood glucose levels using the glucometer provided. The first exercise session will consist of a 40-minute treadmill walk/jog at ~40-50% of VO2max. The second exercise session will include various aerobic and anaerobic activities including push-ups, plank, jumping jacks, high knees, etc. Regular finger capillary blood samples will be collected every 10-minutes during exercise. Once the exercise session is complete, participants will be asked to remain in the laboratory for 30-minutes for additional blood glucose measurements and to ensure hypoglycemic episodes do not occur post-exercise. Participants will be given the contour link glucometer to monitor glucose levels throughout the evening and night.

ELIGIBILITY:
Inclusion Criteria:

* Have had diabetes for > 1 year
* Currently treated with continuous subcutaneous insulin infusion (CSII)/insulin pump therapy for at least 6 months
* Fair-to-good glycemic control (last HbA1c ≤ 9.0%)

Exclusion Criteria:

* Frequent and unpredictable hypoglycemia
* Unable to exercise on a regular basis due to an injury or other restriction
* Using an insulin pump and switch to injections (or vice versa) in the last two months
* Have conditions that would make exercise unsafe (e.g. high blood pressure)
* Take medications in the class of drugs called 'beta-blockers'
* A woman who is pregnant, planning pregnancy, or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants were recruited by random sampling as well as an email blast using previous studies that involved individuals with type 1 diabetes on insulin pump therapy and regularly active. The previous research project at York University had the same inclusion criteria, so that email list will be used to contact those individuals for this study as well.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Blood glucose concentrations | Approximately 2 hours
  Whole blood glucose concentrations were measured using a handheld glucometer every 10-minutes before, during, and after both exercise conditions.

SECONDARY OUTCOMES:
Participants estimated blood glucose concentration | 40-minutes during exercise and 10-minutes post-exercise
  Whole blood glucose concentrations were measured using a handheld glucometer and the values were blinded from participants during exercise. Participants were asked to estimate the change in glycemia every 10-minutes and actual measured blood glucose was revealed to participants post-exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Riddell, PhD, Principal Investigator — York University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iscoe KE, Riddell MC. Continuous moderate-intensity exercise with or without intermittent high-intensity work: effects on acute and late glycaemia in athletes with Type 1 diabetes mellitus. Diabet Med. 2011 Jul;28(7):824-32. doi: 10.1111/j.1464-5491.2011.03274.x. PMID 21388440
- [Result] Guelfi KJ, Ratnam N, Smythe GA, Jones TW, Fournier PA. Effect of intermittent high-intensity compared with continuous moderate exercise on glucose production and utilization in individuals with type 1 diabetes. Am J Physiol Endocrinol Metab. 2007 Mar;292(3):E865-70. doi: 10.1152/ajpendo.00533.2006. PMID 17339500
- [Result] Yardley JE, Sigal RJ. Exercise strategies for hypoglycemia prevention in individuals with type 1 diabetes. Diabetes Spectr. 2015 Jan;28(1):32-8. doi: 10.2337/diaspect.28.1.32. PMID 25717276